#### NCT03181009

Full Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Immune Markers after Minimum Maintenance Dose

Short Title: Multi Immunotherapy to test Minimum dose using Xolair (MIMiX)

Informed Consent – Approval Date: June 12, 2018

Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Immune Markers after Minimum Maintenance Dose

Please check all that are applicable:

I am an adult participant in this study.

Print your name here:

I am the parent or guardian granting permission for a child in this study (the use of "you" refers to "your child" or "your ward.")

Print child's name here:

\*\*\*\*\*\*\*\*\*\*\*\*

Are you participating in any other research studies? \_\_\_\_\_ Yes \_\_\_\_\_No

#### **PURPOSE OF RESEARCH**

You are invited to participate in a research study to test the safety and efficacy of Oral ImmunoTherapy (OIT) with omalizumab (Xolair, anti-IgE) to help children and adults who are allergic to food be able to safely tolerate food allergens. Specifically in this protocol, the food allergens will include at least two, maximum of five of the following: peanut, almond, cashew, walnut, hazelnut, milk, egg, wheat, soy, sesame seed, cod, shrimp, and/or salmon. Omalizumab is considered an investigational drug for the treatment of food allergies in children and adults. Investigational means it has not been approved by the Food and Drug Administration (FDA) for use in food allergies in the U.S.

The purpose of this study is to test whether omalizumab improves the safety of OIT, and if omalizumab treatment with multiple food allergen OIT allows the use of a lower maintenance dose of each food allergen in the OIT regimen, particularly in younger subjects with food allergies.






Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

You are being asked to participate in this experimental research study because you have a history of multiple food allergies.

If you decide to terminate your participation in this study, you should notify the Protocol Director, Dr. Kari Nadeau or the co-Protocol Director Dr. Sayantani Sindher at (650) 724-0293.

This research study is looking for 60 participants, between 2 and 25 years of age, with multiple food allergies. Enrollment will occur at 2 centers in the United States. Sean N Parker Center for Allergy and Asthma Research at Stanford University expects to enroll approximately 30 research study participants.

#### **VOLUNTARY PARTICIPATION**

Your participation in this study is entirely voluntary. Your decision not to participate will not have any negative effect on you or your medical care. You can decide to participate now, but withdraw your consent later and stop being in the study without any loss of benefits or medical care to which you are entitled.

#### **DURATION OF STUDY INVOLVEMENT**

This research study is expected to take approximately 26 weeks:

- About 1 day for screening
- 8 weeks for omalizumab administration
- 18 weeks of oral desensitization therapy

#### **PROCEDURES**

If you choose to participate, Dr. Kari Nadeau, Dr. Sayantani Sindher and/or the research study staff will explain the study to you and ask you to read this consent form. The study personnel will answer any questions you may have about the study and what is being asked of you. If you decide to participate you will be asked to sign this consent form and a copy will be given to you.

While participating in this study, you must be very careful to avoid all allergens apart from what is instructed by Dr. Kari Nadeau/Sayantani Sindher and her team during the study, as this may potentially cause an allergic reaction. Also, you may not change your diet or add new foods during your participation in this study.

There will be at least 9 visits to the clinic throughout the study. The study includes:


Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Immune Markers after Minimum Maintenance Dose

- Screening Visit (within 30 days of 1st Omalizumab dose)
- Omalizumab Administration Visits (3 doses 4 weeks apart)
- Build Up (start after last Omalizumab dose until 8 weeks post Omalizumab)
- Maintenance (over 10 weeks)
- End of Study

All participants will receive omalizumab as a subcutenous (under the skin) injection thrice over 8 weeks (at week -8, -4 and week 0) with 4 week intervals between injections. Your specific allergens will be introduced in an oral desensitization day at week 0, after the last dose of omalizumab. You will be randomly assigned to build up your dose of 300mg or 1200mg daily. There is a 50% chance you will be assigned to either group. Each daily food flour dose will contain about the same amount of each allergen protein composed of 2-5 of your allergens. You will increase your allergen dose to reach the goal of a maintenance dose 300mg or 1200mg every day, depending on which group you are assigned, without having an allergic reaction. The amount of time to reach this will be about 8 weeks. Oat flour may be added to your daily food flour dose in order to ensure that neither you nor the study team knows to which arm you are assigned (double blind). Once the goal dose is reached, you will continue to take the same food flour doses daily until week 18.

#### Baseline/Screening Visit

We will ask you to come first for a screening visit to perform procedures to determine if you are eligible for the study, and to review your medical history regarding your food allergies, other allergies and general health. We may ask to contact your primary provider or allergist to get a copy of any medical records pertaining to your food allergies.

At this screening visit, the following procedures will be performed after you sign this informed consent form:

- Review of medical history
- Physical examination (including height and weight)
- Vital signs (heart rate, respiratory rate, temperature, and blood pressure)
- Spirometry (a test that uses a hand held instrument connected to a computer to measure how deep a breath you can take and how fast you can blow air out through your mouth) or Peak Flow Meter (a small tube with a mouthpiece that measures how fast you can blow air out through your mouth) reading,
- Skin prick test may be done to assess your sensitivity to food allergens. You may be asked to stop taking antihistamines such as Benadryl, Zyrtec, or Claritin, before the visit in order to undergo a skin prick test.






Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

- Review of medications you are currently taking
- Urine pregnancy test for female patients of childbearing potential. Your urine samples will be destroyed right after the laboratory tests are completed.
- Blood draw (not more than 50mL or 3-4 tablespoons in volume) for foodspecific Immunoglobulins (IgE and IgG4) and for mechanistic studies/immunology markers
- Review of eligibility: you must have food specific IgE>4kU/L in the blood for each allergen OR a skin test reactivity to each food allergen greater than or equal to 6mm wheal diameter for at least two allergens.
- Training on the following will be done at screening and at each subsequent study visit:
  - How to properly store and administer the study dose
  - How to recognize allergic reactions and/or other adverse events
  - o What actions you must take should you have an allergic reaction
  - How and when to use the epinephrine-containing autoinjector. You and/or your families will be required to have an epinephrine autoinjector with you at all times. If you do not have the auto injector, you will be given a prescription for an epinephrine-containing autoinjector (EpiPen Jr. or EpiPen) at the beginning of the study.

The visit will be approximately 2-3 hours long

#### Omalizumab Administration Visits - Week -8 and Week -4

At week -8 visit, if you continue to be eligible for the study, you will receive your first dose of omalizumab as a subcutaneous (under the skin) injection at this visit. Your second dose of Omalizumab will be administered at week-4 visit. Each time omalizumab is administered, you will be closely observed at the clinic for approximately  $1 \frac{1}{2}$  hours after the injection.

A symptom directed physical exam, review of medications and any change in your health will be performed at these visits.

Each visit will be at least 2 hours long.

#### Oral Immunotherapy - Week 0

At week 0 visit, you will receive your last omalizumab dose. You will also begin oral desensitization with 5mg total protein dose of 2 to 5 foods you are allergic to. You will take your first oral dose 1 hour after the omalizumab injection.

After the 5 mg dose, you will be observed for a minimum of 2 hours in clinic. Physical Exam, serial vital signs, review of medications and any health change, and spirometry will be performed at this visit.

You will also be instructed to keep a daily electronic diary to document that you have taken your daily dose and any symptoms that occur at home.






Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

If you do not tolerate 5mg total protein of your allergens, you will be asked to leave the study.

If you are able to tolerate the 5 mg dose, you will be given your allergen doses to take at home. You will take your food flour dose every day. Dosing instructions will be provided, including a 24-hour emergency contact information and contact information for the research team.

You will also be instructed to keep a daily electronic diary to document that you have taken your daily dose and any symptoms that occur at home.

The food allergy action plan and epinephrine auto injector use will also be reviewed.

#### Oral Immunotherapy- Week 4 through 16

You will increase your allergen dose to reach the goal of a maintenance dose 300mg or 1200mg every day, depending on which group you are assigned. Once the dose is reached, you will remain at the same daily dose until week 18.

At each new dose, you will take the first dose in the clinic followed by an observation period of a minimum of 2 hours.

You will continue to take daily food flour dose at home unless advised otherwise by the study doctor or designee. You will be asked to return to the clinic every 4 weeks to have the dose increased as appropriate. The study doctor may ask you to come in sooner than 4 weeks in order to assess how you are doing, and possibly adjust the allergen dose if necessary.

At each visit, physical exam, serial vital signs, review of medications and any health change, spirometry, and diary review will be performed.

The food allergy action plan and epinephrine auto injector use will also be reviewed.

#### End of Active Phase of Study (Week 18)

The following will be completed at the end of study visit or if you prematurely discontinue from the study:

- Physical examination (including height and weight)
- Vital signs
- Spirometry (a test that uses a hand held instrument connected to a computer to measure how deep a breath you can take and how fast you can blow air out through your mouth) or Peak Flow Meter (a small tube with a mouthpiece that measures how fast you can blow air out through your mouth) reading,
- Skin prick testing. You may be asked to stop taking antihistamines such as Benadryl, Zyrtec, or Claritin, before the visit




Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Immune Markers after Minimum Maintenance Dose

- Review of medications you are currently taking

- Urine pregnancy test for female patients of childbearing potential. Your urine samples will be destroyed right after the laboratory tests are completed.
- Blood draw (not more than 50mL or 3-4 tablespoons in volume) for foodspecific Immunoglobulins (IgE and IgG4) and for mechanistic studies/immunology markers
- Review of food allergy action plan and epinephrine auto injector use

#### Throughout the study

- You will keep electronic diaries during the study to document that you have taken your dose and any symptoms that occur at home.
- You will be asked to continue to follow a food elimination diet of your food allergens and will be continually monitored for compliance by thorough questioning and review of the electronic diaries at every study clinic visit.
- If you miss any of your food flour doses, you will be asked to inform the study team and ask for guidance on how to proceed with dosing.
- You will be asked to bring all unused allergen dose(s) at every clinic visit.

#### Women of Childbearing Potential

If you are pregnant or currently breast feeding, you may not participate in this study since the risk of omalizumab to a developing fetus or breastfeeding child is currently unknown and could be potentially dangerous.

If you are a woman of childbearing potential, it is expected that you will use an effective method of birth control to prevent exposing a fetus to a potentially dangerous agent with unknown risk.

To confirm to the extent medically possible that you are not pregnant, you agree to have a pregnancy test done at screening and prior to starting omalizumab therapy. You must agree to avoid sexual intercourse or use a birth control method judged to be effective by the investigator and which will not interfere with the proposed investigation. You must accept the risk that pregnancy could still result despite the responsible use of reliable method of birth control. You agree to notify the investigator as soon as possible of any failure of proper use of your birth control method, or if you become pregnant, either of which may result in your being withdrawn from the study.

#### Tissue Sampling for Research

Research using tissues (blood) is an important way to try to understand human disease. You have been given this information because the investigators want to






STUDY

Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

include your blood in a research project and because they want to save the samples for future research. There are several things you should know before allowing your tissues to be studied.

Your blood sample will be stored for an indefinite period of time under a unique numbered identifier in the Nadeau Research lab. Your samples will be sent outside of Stanford University for analysis. These research studies are very important to understand the changes in the immune system that may occur as you become desensitized to your allergens. These results may help us to design better treatments in the future for multi food allergic patients.

You have the right to refuse to allow your tissues to be studied now or saved for future study. You may withdraw from this study at any time. The investigators might retain the identified samples, e.g., as part of your routine clinical care, but not for additional research.

The results of the study of your samples will be used for research purposes only and you will not be told the results of the tests.

| I consent to my samples being saved for future research | |
|----------------------------------------------------------------|----|
| I do not consent to my samples being saved for future research | :h |

#### PARTICIPANT RESPONSIBILITIES

As a participant, your responsibilities include:

- Follow the instructions of the study doctor and study staff.
- Take the study drug daily as instructed.
- Call the 24/7 on call number if you missed any doses or have any allergic reactions.
- Keep your study appointments. If it is necessary to miss an appointment, please contact the study doctor or research study staff to reschedule as soon as you know you will miss the appointment.
- Tell the study doctor or research study staff about any side effects, doctor visits, or hospitalizations that you may have.
- Tell the study doctor or research staff if you believe you might be pregnant or gotten your partner pregnant.
- Keep the study drug in a safe place, away from children and for your use only.


Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Immune Markers after Minimum Maintenance Dose

- Keep your electronic diaries as instructed.
- Ask questions as you think of them.
- Tell the study doctor or research staff if you change your mind about staying in the study.

#### WITHDRAWAL FROM STUDY

If you first agree to participate and then you change your mind, you are free to withdraw your consent and discontinue your participation at any time. Your decision will not affect your ability to receive medical care for your disease and you will not lose any benefits to which you would otherwise be entitled.

If you decide to withdraw your consent to participate in this study, you should notify the Protocol Director Dr. Kari Nadeau or the co-Protocol Director Sayantani Sindher at (650) 724-0293.

If you withdraw from the study, or the study medication is stopped for any reason,

- You will be asked to return to clinic for an end of study visit
- You must return all study-related supplies, including unused study drug.

The study doctor may also withdraw you from the study and the study medication may be stopped, without your consent for one or more of the following reasons:

- Failure to follow the instructions of the investigator and study staff.
- The Investigator decides that continuing your participation could be harmful to you (including psychological and/or emotional strains).
- Pregnancy
- You need treatment not allowed in the study.
- The study is cancelled.
- Other administrative reasons.
- Unanticipated circumstances.

### POSSIBLE RISKS, DISCOMFORTS, AND INCONVENIENCES

There are risks, discomforts, and inconveniences associated with any research study. These deserve careful thought. You should talk with the study investigator if you have any questions.

The potential discomforts with the desensitization procedure and OIT may include an itchy rash, hives, nausea, abdominal discomfort, vomiting, diarrhea, facial swelling, cough, stuffy, runny nose, sneezing, wheezing, and shortness of breath.


Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

The major risks involved include severe breathing difficulties and rarely anaphylactic shock (severe allergic reaction involving many of the above symptoms plus sudden drop in blood pressure and loss of consciousness). A severe allergic reaction would require immediate medical treatment and could result in permanent disability or death. Medication, personnel, and equipment will be immediately available to treat allergic reactions. You will also be provided a prescription for an Epinephrine autoinjector to have with you at all times and to use in case of an allergic reaction.

The other major concern besides anaphylaxis is eosinophilic esophagitis (EoE). EoE is a condition where a type of white blood cell (eosinophil) builds up in the tube that connects your mouth to your stomach (esophagus). This can cause stomach/chest pain, vomiting, regurgitation, and/or difficulty swallowing. It is possible that EoE may be reversed upon stopping dosing.

The risk involved with skin testing includes discomfort from the needle prick, along with itching and swelling at the skin test site in positive responses. Less common side effects include severe allergic reactions. You may be given topical steroid creams for application to the affected areas if needed.

Risks with blood draws include fainting, local pain, stinging, bleeding, or bruising at the site where the needle is inserted into the vein. On rare occasions infection at the needle stick site may occur.

#### **Omalizumab Risks**

Omalizumab is approved by the FDA for patients aged 6 years and older with moderate to severe asthma.

The adverse event profile (bad side effects) of omalizumab observed during the clinical development program was very similar to placebo with the most commonly reported adverse reactions being mild reactions at the place on the skin where the omalizumab was injected (injection site reactions). The overall frequency of injection site reactions was similar in omalizumab-treated patients and placebo patients. Other than injection site reaction, the most frequently reported adverse events were nasopharyngitis, upper respiratory tract infection and headache. During clinical studies with adult and adolescent patients 12 years of age and older, the most commonly reported adverse reactions were injection site reactions, including injection site pain, swelling, erythema (redness), pruritus (itching) and headaches. In clinical studies with patients 6 to <12 years of age, the most commonly reported adverse reactions were headache, pyrexia (fever) and upper abdominal pain. Most of the adverse events were mild or moderate in severity.


Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

Here is the list of the adverse reactions recorded in clinical studies in the total allergic asthma safety population and in patients with chronic spontaneous/idiopathic urticaria (CSU/CIU) treated with omalizumab:

- Very common (≥1/10): pyrexia (fever), headache
- Common (>1/100; <1/10): headache, upper abdominal pain, injection site reactions such as pain, erythema (redness), pruritus (itching), and swelling, nasopharyngitis (inflammation of the nose and throat), sinusitis, viral upper respiratory tract infection, arthralgia (joint pain)
- Uncommon (>1/1000; <1/100): pharyngitis (throat swelling), dizziness, somnolence (sleepiness), paresthesia (tingling, numbness, or burning), syncope (fainting), postural hypotension, flushing, coughing, allergic bronchospasm, nausea, diarrhea, dyspeptic signs and symptoms (upset stomach), urticaria (hives), rash, pruritus (itching), photosensitivity, weight increase, fatigue, swelling arms, influenza-like illness</li>
- Rare (<1/1000): parasitic infections, anaphylactic reaction and other allergic conditions, anti- therapeutic antibody development, laryngoedema (throat swelling), angioedema (swelling)

Additional events reported in CSU/CIU studies with incidence  $\geq 1\%$  in any treatment group and  $\geq 2\%$  higher in any omalizumab group than placebo: toothache, upper respiratory tract infections, urinary tract infection, fungal infection, sinus headache, myalgia, pain in extremity, musculoskeletal pain, fever, and injection site reactions occurred during the studies in more omalizumab -treated patients than placebo patients.

The listing of adverse reactions from post-marketing spontaneous reports (mostly from patients with asthma) include:

- Immune system disorders: Anaphylaxis and anaphylactoid reactions have been reported following the first or subsequent administrations, serum sickness
- Skin and subcutaneous disorders: Alopecia (hair loss)
- Blood and lymphatic system disorders: Idiopathic severe thrombocytopenia (decrease of platelets)
- Arterial thromboembolic events (ATEs) included stroke, transient ischemic attack, myocardial infarction, unstable angina, and cardiovascular death (including death from unknown cause)
- Respiratory, thoracic and mediastinal disorders: Allergic granulomatous angiitis (i.e. Churg Strauss syndrome, inflammation of the blood vessels)
- Musculoskeletal and connective tissue disorders: Arthralgia (joint pain), myalgia (muscle pain), joint swelling






Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Immune Markers after Minimum Maintenance Dose

Malignant neoplasms (cancer)

Antibody formation to omalizumab (not associated with any adverse events)

Of the adverse events of special interest, anaphylactic reactions (presenting as wheezing, shortness of breath, cough, chest tightness, or trouble breathing, flushing, itching, hives, or feeling warm, swelling of the throat or tongue, throat tightness, hoarse voice, or trouble swallowing, low blood pressure, dizziness, fainting, rapid or weak heartbeat, anxiety) were observed but were rare and typically occurring within 2 hours of the first injection. Anaphylaxis is a lifethreatening condition and can lead to death. There were no reported cases of anaphylaxis with a fatal outcome in any of the clinical studies. Fatal cases with anaphylaxis have been reported in the post marketing pharmacovigilance reports since 2003. None of these fatal cases with anaphylaxis were due to Xolair.

Cases of cancer were observed in some people who received omalizumab. Although more cases of malignancy (cancers) were observed in the omalizumab treatment group compared with the control group, the short exposure duration is not consistent with the biology of cancer pathogenesis; additionally, the diversity in the type of cancers observed and the clinical features of the individual cases render a causal relationship unlikely. However, study limitations preclude definitively ruling out a malignancy risk with omalizumab.

Some people who received omalizumab have had heart and circulation problems such as chest pain, heart attack, blood clots in the lungs or legs, or temporary symptoms of weakness on one side of the body, slurred speech, or altered vision. It is not known whether this is caused by omalizumab.

Inflammation of the blood vessel rarely happened in people with asthma who received omalizumab. This usually, but not always, happened in people who also take a steroid medicine by mouth that is being stopped or the dose is being lowered. It is not known whether this is caused by omalizumab. Tell your study doctor right away if you have rash, chest pain, shortness of breath, or a feeling of pins and needles or numbness of your arms or legs.

Some people who are at a high risk for parasite (worm) infections, can get a parasite infection after receiving omalizumab. In patients at chronic high risk of helminth (worm) infection, a placebo-controlled trial showed a slight increase in infection rate with omalizumab, although the course, severity, and response to treatment of infection were unaltered. The helminth (worm) infection rate in the overall clinical program, which was not designed to detect such infections, was less


Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

than 1 in 1,000 patients. However, caution may be warranted in people at high risk of helminth infection, in particular when traveling to areas where helminthic infections are endemic.

#### **POTENTIAL BENEFITS**

We cannot and do not guarantee or promise that you will receive any benefits from this study. You may benefit from a decrease in the sensitivity to your allergens, and improve your immune protection to the offending food allergens. The knowledge gained from this study may aid in the advancement and understanding of food allergy and help in the development of new approaches for its treatment or prevention.

#### **ALTERNATIVES**

The alternative to participating is to continue food avoidance, which is standard of treatment for food allergic individuals.

#### **PARTICIPANT'S RIGHTS**

You should not feel obligated to agree to participate. Your questions should be answered clearly and to your satisfaction. If you decide not to participate, tell the study doctor.

You will be told of any important new information that is learned during the course of this research study, which might affect your condition or your willingness to continue participation in this study.

#### ClinicalTrials.gov

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### **CONFIDENTIALITY**

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed except as authorized by you or as required


Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Immune Markers after Minimum Maintenance Dose

by law. However, there is always some risk that even de-identified information might be re-identified.

Patient information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

The purpose of this research study is to obtain data or information on the safety and effectiveness of OIT and omalizumab; the results will be provided to the sponsor, the Food and Drug Administration and other federal and regulatory agencies as required.




Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

# **Authorization To Use Your Health Information For Research Purposes**

Because information about you and your health is personal and private, it generally cannot be used in this research study without your written authorization. If you sign this form, it will provide that authorization. The form is intended to inform you about how your health information will be used or disclosed in the study. Your information will only be used in accordance with this authorization form and the informed consent form and as required or allowed by law. Please read it carefully before signing it.

## What is the purpose of this research study and how will my health information be utilized in the study?

The purpose of this study is to see if using omalizumab can help adults and children with food allergies be able to tolerate those same foods. The study doctor, Dr. Sayantani Sindher and/or Dr. Kari Nadeau, will use your personal health information to complete this research. Regulatory authorities such as the FDA and the IRB may also review or copy your information to make sure that the study is done properly or for other purposes required by law. The results of this study may be published in a medical journal and shown at medical meetings. You will not be identified (by name or any other means) in any of these publications.

## Do I have to sign this authorization form?

You do not have to sign this authorization form. But if you do not, you will not be able to participate in this research study, including receiving any research-related treatment.

Signing the form is not a condition for receiving any medical care outside the study.

If I sign, can I revoke it or withdraw from the research later?


Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

If you decide to participate, you are free to withdraw your authorization regarding the use and disclosure of your health information (and to discontinue any other participation in the study) at any time. After any revocation, your health information will no longer be used or disclosed in the study, except to the extent that the law allows us to continue using your information (e.g., necessary to maintain integrity of research). If you wish to revoke your authorization for the research use or disclosure of your health information in this study, you must write to: Dr. Kari Nadeau or Dr. Sayantani Sindher at 269 Campus Drive, CCSR Building, Room 3215, Stanford, CA 94305, phone number: 650-724-0293

## What Personal Information Will Be Obtained, Used or Disclosed?

Your health information related to this study, may be used or disclosed in connection with this research study, including, but not limited to, your demographic information (including date of birth, gender, race/ethnicity, and medical record number), medical history, history of allergies, physical examinations, lab test results.

## Who May Use or Disclose the Information?

The following parties are authorized to use and/or disclose your health information in connection with this research study:

- The Protocol Director, Dr. Kari Nadeau and the co-Protocol Director Dr. Sayantani Sindher
- The Stanford University Administrative Panel on Human Subjects in Medical Research and any other unit of Stanford University as necessary
- Research Staff

## Who May Receive or Use the Information?

The parties listed in the preceding paragraph may disclose your health information to the following persons and organizations for their use in connection with this research study:




Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

- The Office for Human Research Protections in the U.S. Department of Health and Human Services
- Data Safety Monitoring Board
- The National Institutes of Health (NIH)
- Regeneron/Adelphi Values
- The Food and Drug Administration
- Research collaborators outside of Stanford

Your information may be re-disclosed by the recipients described above, if they are not required by law to protect the privacy of the information.

## When will my authorization expire?

Your authorization for the use and/or disclosure of your health information will end on December 31, 2100 or when the research project ends, whichever is earlier.

## Will access to my medical record be limited during the study?

To maintain the integrity of this research study, you may not have access to any health information developed as part of this study until it is completed. At that point, you would have access to such health information if it was used to make a medical or billing decision about you (e.g., if included in your official medical record).

| Signature of Adult Participant | Date |
|---|---|
| Print Name of Adult Participant | |
| Signature of Legally Authorized Representative (LAR) (e.g., parent, guardian or conservator) | Date |






Approval Date: June 12, 2018 Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Immune Markers after Minimum Maintenance Dose

Print Name of LAR

LAR's Authority to Act for Participant (e.g., parent, guardian or conservator)


Participant ID:



STUDY

Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

#### FINANCIAL CONSIDERATIONS

#### **Payment**

You will not be paid to participate in this research study.

#### Costs

There is no cost to you for participating in this study, other than basic expenses like transportation and the personal time it will take to come to all of the study visits.

#### **Sponsor**

This study is being funded by private funding sources, the National Institutes of Health (NIH), and by Regeneron/Adelphi Values.

#### COMPENSATION for Research-Related Injury

All forms of medical diagnosis and treatment – whether routine or experimental – involve some risk of injury. In spite of all precautions, you might develop medical complications from participating in this study. If such complications arise, the Protocol Director and the research study staff will assist you in obtaining appropriate medical treatment. In the event that you have an injury or illness that is directly caused by your participation in this study, reimbursement for all related costs of care first will be sought from your insurer, managed care plan, or other benefits program. You will be responsible for any associated co-payments or deductibles as required by your insurance.

If costs of care related to such an injury are not covered by your insurer, managed care plan or other benefits program, you may be responsible for these costs. If you are unable to pay for such costs, the Protocol Director will assist you in applying for supplemental benefits and explain how to apply for patient financial assistance from the hospital.

You do not waive any liability rights for personal injury by signing this form.

#### **CONTACT INFORMATION**

Questions, Concerns, or Complaints: If you have any questions, concerns or complaints about this research study, its procedures, risks and benefits, or alternative courses of treatment, you should ask the Protocol Director, Dr. Kari Nadeau or the co-Protocol Director Dr. Sayantani Sindher at (650) 724-0293. You


Participant ID:



STUDY

Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test

Immune Markers after Minimum Maintenance Dose

should also contact her at any time if you feel you have been hurt by being a part of this study.

Independent Contact: If you are not satisfied with how this study is being conducted, or if you have any concerns, complaints, or general questions about the research or your rights as a participant, please contact the Stanford Institutional Review Board (IRB) to speak to someone independent of the research team at (650)-723-5244 or toll free at 1-866-680-2906. You can also write to the Stanford IRB, Stanford University, 3000 El Camino Real, Five Palo Alto Square, 4th Floor, Palo Alto, CA 94306.

Appointment Contact: If you need to change your appointment, please contact snpcenterallergy.scheduler@stanford.edu

#### **EXPERIMENTAL SUBJECT'S BILL OF RIGHTS**

As a research participant you have the following rights. These rights include but are not limited to the participant's right to:

- be informed of the nature and purpose of the experiment;
- be given an explanation of the procedures to be followed in the medical experiment, and any drug or device to be utilized;
- be given a description of any attendant discomforts and risks reasonably to be expected;
- be given an explanation of any benefits to the subject reasonably to be expected, if applicable;
- be given a disclosure of any appropriate alternatives, drugs or devices that might be advantageous to the subject, their relative risks and benefits;
- be informed of the avenues of medical treatment, if any available to the subject after the experiment if complications should arise;
- be given an opportunity to ask questions concerning the experiment or the procedures involved;
- be instructed that consent to participate in the medical experiment may be withdrawn at any time and the subject may discontinue participation without prejudice;
- be given a copy of the signed and dated consent form; and
- be given the opportunity to decide to consent or not to consent to a medical experiment without the intervention of any element of force, fraud, deceit, duress, coercion or undue influence on the subject's decision.




Approval Date: June 12, 2018 Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Immune Markers after Minimum Maintenance Dose

| May we contact you about future studies that Yes No | nt may be of intere | est to you? |
|---|---|---|
| Signing your name means you agree to be in copy of this signed and dated consent form. | | nat you will receive a |
| Signature of Adult Participant | | Date |
| Print Name of Adult Participant | _ | |
| Signature of Legally Authorized Representation (e.g., parent, guardian or conservator) | ve (LAR) | Date |
| Print Name of LAR | _ | |
| LAR's Authority to Act for Participant (e.g., parent, guardian or conservator) | _ | |
| (If available) Signature of Other Parent or G | <br>uardian | Date |
| Print Name of Other Parent or Guardian | _ | |
| Authority to Act for Participant | _ | |






Approval Date: <u>June 12, 2018</u> Expiration Date: April 11, 2019

#### STANFORD UNIVERSITY Research Consent Form

Protocol Director: Kari Nadeau, MD PhD

Protocol Title: A Phase 2 Study of Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Immune Markers after Minimum Maintenance Dose

The IRB determined that the permission of two parents is recommended in accordance with 21 CFR 50.55 unless one parent is deceased, unknown, incompetent, not reasonably available, or only one parent has legal responsibility for the care and custody of the child. *Not reasonably available* means that the other parent is not present during the consenting process, or will not be available prior to the start of research procedures.

| Signature of Person Obtaining Consent | Date |
|----------------------------------------|------|
| Print Name of Person Obtaining Consent | |






Consent V3 07 May 2018